CLINICAL TRIAL: NCT04936243
Title: A Randomized Control Trial of Telemedicine vs In Person Oncology Patient Surveillance
Brief Title: TIPOPS (Telemedicine vs In Person Oncology Patient Surveillance)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christopher Manz, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-192
Record Dates: First submitted 2021-06-18; First posted 2021-06-23 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Prostate Cancer; Patient Engagement; Patient Preference; Patient Satisfaction
Keywords: Breast Cancer; Prostate Cancer; Patient Engagement; Patient Preference; Patient Satisfaction
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Patient Participation; Patient Preference; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLLOW UP VISIT-TELEMEDICINE (Experimental): After initial in-person routine followup care, participants will be randomly assigned to receive telemedicine care delivery for their subsequent follow up appointment. Participants will complete a survey after each visit.
  Interventions: Behavioral: FOLLOW UP VISIT-TELEMEDICINE
- FOLLOW UP VISIT-FACE TO FACE (Experimental): After initial in-person routine followup care, participants will be randomly assigned to receive face-to-face care delivery for their subsequent follow up appointment. Participants will complete a survey after each visit.
  Interventions: Behavioral: FOLLOW UP VISIT-FACE TO FACE

INTERVENTIONS:
Behavioral: FOLLOW UP VISIT-TELEMEDICINE — Routine follow up care conducted remotely with video-conferencing tools
  Arms: FOLLOW UP VISIT-TELEMEDICINE
Behavioral: FOLLOW UP VISIT-FACE TO FACE — Routine follow up care conducted in person
  Arms: FOLLOW UP VISIT-FACE TO FACE

SUMMARY:
This research study is comparing telemedicine and face-to-face visits to understand patients' experiences with telemedicine versus face to face visits and to understand when it is and is not appropriate to conduct visits remotely

DETAILED DESCRIPTION:
This study is a prospective randomized trial of telemedicine (TM) versus face-to-face (F2F) visits for follow up care of patients with either early-stage breast or prostate cancer.

This study does not involve investigational drugs or devices but does involve survey data collection from participants about their experiences of care.

After an initial in-person routine visit, participants will be randomly assigned to either telemedicine or face-to-face care delivery for their next routine visit.

It is anticipated participants will be in the study for about 6 months depending on the timing of their routine care appointments.

It is expected that 360 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* For breast cancer participants: Early-stage breast cancer defined as Stages I-IIIA at diagnosis or localized prostate cancer defined as Stages I-III
* For breast cancer participants: participant has completed definitive treatment for early stage breast cancer including surgery, radiation, chemotherapy, anti-HER2 antibody treatment. Participant may or may not be taking oral anti-estrogen treatment such as tamoxifen or an aromatase inhibitor
* For prostate cancer participants: participant is on active surveillance or has undergone definitive surgery for localized prostate cancer
* Participant is on a surveillance follow up visit schedule occurring at every three to seven month intervals
* Willingness and ability to use Patient Gateway portal
* Participant has access to an electronic device that can support a video and audio virtual visit platform (for example, laptop computer, desktop computer, smart phone)
* Participants can be women or men
* Age ≥ 18 years

Exclusion Criteria:

* Patients whose next visit requires cytotoxic chemotherapy, radiation therapy, anti-HER2 antibody therapy or investigational cancer agents are ineligible
* Patients with distant metastatic breast cancer
* Patients with locally advanced or metastatic prostate cancer
* Patients treated by radiation therapy for prostate cancer
* Patients whose next visit requires a prostate biopsy
* Prisoners
* Non-English speaking patients (non-English speaking patients will be excluded from the trial given the challenges of delivering telemedicine with the use of medical interpreters. There are also logistical challenges in obtaining the study endpoints, which are largely survey based, with non-English speakers as well as the possibility that study endpoints will be influenced by the presence of a medical interpreter during a visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Patient Experience Comparison | Up to 6 months
  Compare early-stage breast and early stage prostate cancer patients' experiences with a one-time Telemedicine (TM) versus Face to Face (F2F) follow up visit for routine oncologic surveillance

SECONDARY OUTCOMES:
Patient preference Comparison | Up to 6 months
  Compare patient preferences for Telemedicine (TM) versus Face to Face (F2F) visits for ongoing cancer care
Indirect Health Care Costs Comparison | Up to 6 months
  Compare patient reported indirect healthcare costs for Telemedicine (TM) versus Face to Face (F2F) follow up visits:
Health system use Comparison | Two weeks after study visit
  Compare participant health system use relating to cancer diagnosis within two weeks after study visit
Clinician Experience Comparison | Up to 6 months
  Compare the clinician experience with Telemedicine (TM) versus Face to Face (F2F) for a one-time surveillance follow up visit for breast or prostate cancer care
Clinician Preference | Up to 6 months
  Assessing clinician preference regarding the appropriate use of telemedicine visits for the follow-up of early stage cancer patients who have completed early active therapy (e.g., surgery, radiation and/or chemotherapy) or are under surveillance
Symptom severity-prostate cancer patients Comparison | Up to 6 months
  Compare patient reported erectile dysfunction and urinary symptoms after undergoing radical prostatectomy between patients who have a TM follow up visit vs. a F2F follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Manz, MD, MSHP, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu